CLINICAL TRIAL: NCT01813006
Title: Effect of Omega-3 Polyunsaturated Fat on Endothelial Function and Inflammatory Parameters in Familial Hypercholesterolemia - a Double Blind, Placebo-controlled Crossover Study
Brief Title: Effect of Omega-3 Fatty Acid on Endothelial Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/899(REK); 2012-000505-68 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2013-03

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Docosahexaenoic Acids; Omacor; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Active Comparator): Omega-3 fatty acids
  Interventions: Drug: Omega-3
- Placebo (Placebo Comparator): Placebo/olive oil
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Omega-3
  Other Names: Omacor
  Arms: Omega-3
Drug: placebo
  Other Names: olive oil
  Arms: Placebo

SUMMARY:
Background

Familial hypercholesterolemia (FH) is an inherited disease in which the level of bad cholesterol (LDL-cholesterol) is increased, leading to an increase in coronary heart disease even if adequately treated with cholesterol lowering medication (statins). Polyunsaturated fatty acids (PUFA) including omega-3 is known to affect the risk for coronary disease, however its effect on patients with FH is not known.

The purpose of the study is to assess the effect of PUFA on patients with FH, with regard to inflammation measured in the blood and the effect on the blood vessels'ability to relax (endothelial function) by means of tonometry.

Hypothesis

Treatment with 4 grams of PUFA a day for 4 months will lead to an improvement in the endothelial function, and the treatment will also lead to a decrease in in several markers of inflammation and in lipids in the blood.

ELIGIBILITY:
Inclusion Criteria:

* documented familial hypercholesterolemia
* age 18-60 years
* on statin treatment for at least 12 months

Exclusion Criteria:

* pregnancy or planned pregnancy
* breast feeding
* cancer
* non-compliance
* PUFA/omega-3 < 3 months before inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | Baseline
  Reactive Hyperemia Index (RHI) is a measure for endothelial function by means of tonometry
Reactive Hyperemia Index (RHI) | 3 months
  Measure of endothelial function
Reactive Hyperemia Index (RHI) | 6 months
  Measure of endothelial function
Reactive Hyperemia Index (RHI) | 9 months
  Measure of endothelial function

SECONDARY OUTCOMES:
Markers of inflammation | Baseline
  Serological markers of inflammation including cytokines, C-reactive protein (CRP) and complement factors
Inflammatory markers | 3 months
  Serological markers of inflammation including cytokines, CRP and complement factors
Inflammatory markers | 6 months
  Serological markers of inflammation including cytokines, CRP and complement factors
Inflammatory markers | 9 months
  Serological markers of inflammation including cytokines, CRP and complement factors

OTHER OUTCOMES:
Lipid parameters | Baseline
  Different fractions of lipids in the blood including LDL-cholesterol, HDL cholesterol, triglycerides and their subfractions
Lipid parameters | 3 months
  Different fractions of lipids in the blood including LDL-cholesterol, HDL cholesterol, triglycerides and their subfractions
Lipid parameters | 6 months
  Different fractions of lipids in the blood including LDL-cholesterol, HDL cholesterol, triglycerides and their subfractions
Lipid parameters | 9 months
  Different fractions of lipids in the blood including LDL-cholesterol, HDL cholesterol, triglycerides and their subfractions

CONTACTS AND LOCATIONS:
Overall Officials: Knut T Lappegård, MD, PhD, Principal Investigator — Nordland Hospital
Locations (1):
- Division of Internal Medicine, Nordland Hospital, Bodø, Norway

REFERENCES:
- [Derived] Hande LN, Thunhaug H, Ludviksen J, Hovland A, Lappegard KT. No effect of omega-3 polyunsaturated fatty acid supplementation on inflammatory markers in familial hypercholesterolemia: a randomized crossover trial. Scand J Clin Lab Invest. 2023 May;83(3):152-159. doi: 10.1080/00365513.2023.2178499. Epub 2023 Mar 31. PMID 36999528